CLINICAL TRIAL: NCT03123952
Title: Expanded Access to ABT-414
Status: No longer available | Type: Expanded Access
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: C16-478; C19-919 (Other: AbbVie)
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Glioblastoma or Solid Tumors, Epidermal Growth Factor Receptor (EGFR) Diagnosis
Keywords: Expanded Access; Pre-approval Access; Compassionate Use; Special Access Program; Named Patient Basis; Special Access Scheme
MeSH Terms: conditions — Glioblastoma; Disease | interventions — ABT-414

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Drug: ABT-414 — ABT-414 will be administered by intravenous infusion

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to ABT-414 prior to approval by the local regulatory agency. Availability will depend on territory eligibility. Participating sites will be added as they apply for and are approved for the EAP. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have epidermal growth factor receptor (EGFR) amplification or EGFRvIII mutation.
* Health Care Provider (HCP) must have prior clinical trial experience with ABT-414.
* The participant must not be eligible for an ABT-414 clinical trial.
* Pediatric participants may be evaluated on a case by case basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie